CLINICAL TRIAL: NCT07389525
Title: Assessment of Drug-Drug Interactions Between Immune Checkpoint Inhibitors and Cytochrome P450 Substrates: Immune Checkpoint Inhibitor (ICI)-Drug-Drug Interaction (DDI) Study
Brief Title: Immune Checkpoint Inhibitor (ICI)-Drug-Drug Interaction (DDI) Study
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Tyler Andrew Shugg, Assistant Professor, Indiana University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: PHARM-IUSCCC-0938
Record Dates: First submitted 2026-01-29; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Gastrointestinal Neoplasms; Genitourinary Cancer; Thoracic Cancer; Sarcoma; Melanoma
Keywords: cytokines; immune checkpoint inhibitor
MeSH Terms: conditions — Gastrointestinal Neoplasms; Urogenital Neoplasms; Sarcoma; Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): CYP enzyme/drug transporter probe substrates administered at two study visits: one before initiation of ICI therapy and one while on therapy.
  Interventions: Drug: ICI Therapy
- Cohort 2 (Experimental): CYP enzyme/drug transporter probe substrates administered at one study visit: during ICI therapy.
  Interventions: Drug: ICI Therapy

INTERVENTIONS:
Drug: ICI Therapy — Low dose of a cocktail of probe substrates for eight major CYP enzymes/drug transporters.

SUMMARY:
Immune checkpoint inhibitors (ICIs) (also called "immunotherapy") are an effective family of anti-cancer drugs, but they can cause serious side effects. Some evidence suggests these side effects might happen because ICIs interact with other drugs that you may already be taking, making those drugs work differently, or causing more side effects. The purpose of this study is to see whether ICIs impact how the liver processes other drugs. To do this, participants will be given a probe cocktail of 7 different FDA-approved drugs that are processed in different ways in the liver.

DETAILED DESCRIPTION:
Findings suggest that adverse events during checkpoint inhibitor therapy may, in part, be caused by drug-drug interactions that increase the risk of adverse events with co-administered medications. Identifying these novel drug-drug interactions will likely inform clinical strategies to reduce adverse events during checkpoint inhibitor therapy and enhance their clinical benefits.

This current research aims to systematically explore the impact of ICIs on CYP/transporter function and the associated risks for adverse events, thereby informing clinical strategies to mitigate these risks and optimize the therapeutic benefits of checkpoint inhibitors. By employing a rigorous crossover drug-drug interaction design, this study seeks to enhance understanding of drug interactions during ICI therapy, ultimately improving patient outcomes in oncology.

The long-term goal of this research is to find ways to manage adverse events that occur during treatment with ICIs. The research has two main aims:

1. To understand how ICI therapy affects the metabolism of certain drugs named CYP/transporter probe drugs and to also understand the risk of side effects from commonly prescribed drugs that are affected by these enzymes and transporters in cancer patients.
2. To examine the relationship between levels of pro-inflammatory cytokines (signaling molecules involved in inflammation) and how well these probe drugs are metabolized before and during ICI therapy.

A two-phase clinical study will be conducted to achieve these aims: patients will be given seven different probe drugs that interact with key enzymes and transporters (CYP1A2, CYP2B6, CYP2C9, CYP2C19, CYP2D6, CYP3A, BCRP, and SLCO1B1) both before they start ICI treatment and after they have begun therapy.

Adverse events will be assessed by looking at how changes in the function of these enzymes and transporters affect the metabolism of drugs that cancer patients commonly use. Special computer models, known as physiologically-based pharmacokinetic (PBPK) models, will be used to simulate how these drugs behave in the body and predict potential serious adverse events.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old at the time of informed consent
* Diagnosed with cancer AND initiating therapy with single agent or combination therapy that includes an immune checkpoint inhibitor (e.g., atezolizumab, cemiplimab, durvalumab, ipilimumab, nivolumab, pembrolizumab, relatlimab, tremelimumab)
* Ability to provide written informed consent and HIPAA authorization

Exclusion Criteria:

* Actively pregnant or breastfeeding
* Body weight less than 50 kg or a BMI >35
* Low baseline hemoglobin, defined as <10 g/dL

  * Note: if a prospective patient's hemoglobin returns to the normal range, they can be re-screened for trial inclusion)
* Past medical history of chronic liver disease, signs and symptom of liver disease (e.g., jaundice, ascites), or aspartate aminotransferase >96 U/L, alanine aminotransferase > 80 IU/L, alkaline phosphatase >260 U/L, or total bilirubin > 2.6 mg/dL

  * Note: if a prospective patient's liver function tests return to the normal ranges, they can be re-screened for trial inclusion)
* Past medical history of chronic kidney disease, signs and symptom of kidney disease (e.g., decreased urine output, swelling in feet and ankles), or estimated glomerular filtration rate <45 mL/minute/1.73 m2 BSA

  * Note: if a prospective patient's kidney function returns to the normal range, they can be re-screened for trial inclusion)
* Poor performance status that makes it unlikely the patient will complete 3 cycles of immune checkpoint inhibitor (at the treating oncologist's discretion)
* Diagnosis or past medical history of autoimmune disorder, including systemic lupus erythematosus, Crohn's disease, Sjogren's syndrome, multiple sclerosis, type 1 diabetes mellitus, Behcet's disease, and ankylosing spondylitis
* History of intolerance, allergic reaction, or hypersensitivity to any of the study drugs (tizanidine, bupropion, flurbiprofen, omeprazole, dextromethorphan, midazolam, rosuvastatin)
* Current infection requiring medical treatment (note: if a prospective patient's infection resolves, they can be re-screened for trial inclusion)
* Concomitant treatment with systemic immunosuppressant drugs (see Appendix 3 for list)

  * Note: patients may be re-screened for trial eligibility if they discontinue any exclusionary drugs for ≥7 days prior to Study Visit 1
* Concomitant treatment with a CYP/transporter probe cocktail drug or strong inhibitors, inducers, or agents that affect the pharmacokinetics of the relevant CYP enzymes or drug transporters (see Appendix 4 for list)

  * Note: patients may be re-screened for trial eligibility if they discontinue any exclusionary drugs for ≥7 days prior to Study Visit 1
* Are unwilling/unable to avoid drugs of abuse, tobacco products or marijuana, or consuming more than 2 alcoholic drinks per day during the study
* Inability to take oral medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in plasma concentrations from drug exposure during ICI therapy | baseline (before start of ICI therapy) up to day 84
Toxicity concentrations for CYP/transporter substrate drugs in plasma | baseline (day before Cycle 1 start) up to day 84
Pro-inflammatory cytokines and CYP/transporter probe drug concentrations in plasma | baseline (day before Cycle 1 start) up to day 84

SECONDARY OUTCOMES:
Assess associations between T cells populations and CYP/transporter probe drug concentrations | baseline (day before Cycle 1 start) up to day 84
  Peripheral blood mononuclear cells (PBMCs)
Concentrations of endogenous biomarkers | baseline (day before Cycle 1 start) up to day 84
  Plasma or urine
CYP/transporter endogenous biomarker concentrations | baseline (day before Cycle 1 start) up to day 84
  Plasma or urine correlated with plasma concentrations of pro-inflammatory cytokines
Correlation of concentration of population of activated T cells and CYP/transporter endogenous biomarkers | baseline (day before Cycle 1 start) up to day 84
  Plasma or urine
CYP/transporter substrate-related adverse events and immune related (ir) adverse events | Baseline (before starting ICI cycle 1) and study visit 2 (up to day 84)
  assessed through surveys given to participants

CONTACTS AND LOCATIONS:
Overall Officials: Tyler Shugg, MD, Principal Investigator — IUSCCC
Locations (1):
- Indiana University Melvin and Bren Simon Comprehensive Cancer Center, Indianapolis, Indiana, United States